CLINICAL TRIAL: NCT04150497
Title: Open Label Dose-escalation and Dose-expansion Study to Evaluate the Safety, Expansion, Persistence and Clinical Activity of UCART22 (Allogeneic Engineered T-cells Expressing Anti-CD22 Chimeric Antigen Receptor) in Patients With Relapsed or refractoryCD22+ B-cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Phase 1/2 Study of UCART22 in Patients With Relapsed or Refractory CD22+ B-cell Acute Lymphoblastic Leukemia (BALLI-01)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellectis S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCART22_01
Record Dates: First submitted 2019-11-01; First posted 2019-11-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: B-cell Acute Lymphoblastic Leukemia (B-ALL); Relapse/Refractory B-ALL; Universal Chimeric Antigen Receptor T-Cell (UCAR-T) Therapy; Allogeneic; Transcription Activator-Like Effector Nuclease (TALEN®)
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Several tested doses of UCART22 until the Maximum Tolerated Dose (MTD) is identified and establish Recommended Phase 2 Dose (RP2D)
  Dose Expansion: UCART22 administered at the RP2D
  Interventions: Biological: UCART22; Biological: CLLS52

INTERVENTIONS:
Biological: UCART22 — Allogeneic engineered T-cells expressing anti-CD22 Chimeric Antigen Receptor given following a lymphodepleting regimen
Biological: CLLS52 — A monoclonal antibody that recognizes a CD52 antigen
  Other Names: Alemtuzumab

SUMMARY:
This is a first-in-human, open-label, dose escalation and expansion study of UCART22 administered intravenously to patients with relapsed or refractory B-cell acute Lymphoblastic Leukemia (B-ALL). The purpose of this study is to evaluate the safety and clinical activity of UCART22 and determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D)

ELIGIBILITY:
Inclusion Criteria:

* B-ALL blast cells expressing CD22
* Diagnosed with R/R B-ALL
* Prior therapy must include at least one standard chemotherapy regimen and at least one salvage regimen

Exclusion Criteria:

-Prior cellular therapy or investigational cellular or gene therapy within 90 days prior to enrollment

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE/SAE/DLT [Safety and Tolerability] | 24 Months
  Incidence, nature, and severity of adverse events and serious adverse events (SAEs) throughout the study in relation to UCART22 and/or lymphodepletion
Dose escalation part: Occurrence of Dose Limiting Toxicities (DLTs) | Up to D28 post initial UCART22 infusion

SECONDARY OUTCOMES:
Investigator assessed overall response rate according to the Response criteria for Acute Lymphoblastic Leukemia (ALL) | At Day 28, Day 56, Day 84, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21 and Month 24
Duration of Response | From the date of the initial response to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 24
Progression Free Survival | From the first day of study treatment to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 24
Overall Survival | From the first day of study treatment to the date of death from any cause, assessed up to Month 24
Pharmacokinetic (PK) profile/exposure levels of CLLS52 (Alemtuzumab) used during lymphodepletion | Lymphodepletion to Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (19):
- United States (14):
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - Sarah Cannon - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center (MSKCC) David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Sarah Cannon - HCA Research Institute, Nashville, Tennessee
  - Sarah Cannon - St. David's South Austin Medical Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Sarah Cannon - Texas Transplant Institute at Methodist Hospital, San Antonio, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- France (5):
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Hôpital Saint Louis, Unité d'Hématologie Adolescents et Jeunes Adultes Département d'Hématologie, Paris
  - Hôpital Robert Debré - Service d'hémato-immunologie, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - CHU Rennes - Hopital Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No